CLINICAL TRIAL: NCT02342496
Title: Probiotics Against Low Grade Inflammation and Increased Intestinal Permeability in the Elderly.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/3
Record Dates: First submitted 2014-12-18; First posted 2015-01-21 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Low-grade Inflammation; Increased Intestinal Permeability
MeSH Terms: interventions — Exercise; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Powder consisting of maltodextrine, treated to resemble the Active product in appearance and taste.
  Interventions: Dietary Supplement: Placebo
- Active, only probiotics (Active Comparator): Powder consisting of freezedried bacteria at 10 billions cfu/daily dose and maltodextrine, treated to resemble the Active product in appearance and taste.
  Interventions: Dietary Supplement: Active, only probiotics
- Active, blend of berries and probiotics (Active Comparator): Powder consisting of freezedried berries , probiotics at 10 billions cfu/daily dose and maltodextrine.
  Interventions: Dietary Supplement: Active, blend of berries and probiotics

INTERVENTIONS:
Dietary Supplement: Placebo — Powder
  Arms: Placebo
Dietary Supplement: Active, only probiotics — Powder
  Arms: Active, only probiotics
Dietary Supplement: Active, blend of berries and probiotics — Powder
  Arms: Active, blend of berries and probiotics

SUMMARY:
The purpose of this study is to evaluate the ability of a blend of berries and probiotics in reducing low-grade inflammation and intestinal permeability in the elderly. The intervention period is one month. Blood and fecal samples will be collected for analysis at baseline and at the end of the intervention with the aim to analyse possible changes in different parameters at the two timepoints. The participants will also be asked to keep a study diary throughout the study period for the documentation of their intestinal health and as a means for checking compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age >75 years
* CRP 2-10 mg/L
* Ability to fill in a study diary by him/herself

Exclusion Criteria:

* Intake of antibiotic treatment in the last 4 weeks before inclusion into the study.
* Currently on corticosteroid treatment
* Presence of chronic inflammatory disease

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
Reduced intestinal permebility measured as decline in the levels of zonulin in blood samples | All blood markers analysed in the study will be measured at start, before the onset of intervention and 4 weeks later at the end of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Malmo, Sweden

REFERENCES:
- [Derived] Lazou-Ahren I, Bjorklund M, Molin G, Xu J, Onning G, Elmstahl S, Jeppsson B. Probiotic-Reduced Inflammaging in Older Adults: A Randomized, Double-Blind, Placebo-Controlled Trial. Probiotics Antimicrob Proteins. 2025 Oct;17(5):3429-3439. doi: 10.1007/s12602-024-10310-7. Epub 2024 Jun 19. PMID 38896223